CLINICAL TRIAL: NCT06386640
Title: A Holistic Patient-centred Intervention to Improve Outcomes of Older People Living With Frailty and Chronic Heart Failure
Acronym: FIT-HF
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0784
Record Dates: First submitted 2024-04-07; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Heart Failure; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phase 3 participants: Phase 3 participants
  Interventions: Other: Intervention Development

INTERVENTIONS:
Other: Intervention Development — Phase I: Research to inform intervention design, Phase II: Co-design and production of intervention with relevant stakeholders, Phase IIa: Physical activity accelerometer data collection and analysis to develop an individualised rehabilitation programme, Phase III: Pilot and refine the intervention across to two NHS sites (University Hospitals of Leicester NHS Trust, Portsmouth Hospitals University NHS Trust).

SUMMARY:
Two-centre complex intervention development and feasibility trial using mixed qualitative and quantitative approach

DETAILED DESCRIPTION:
The intervention will be developed and its effectiveness and feasibility tested via 3 stages: Stage1: Relevant background research will be performed to inform intervention design; stage 2: the intervention will be co-designed with relevant stakeholders and stage 3: the developed intervention will be trialled in a multicentre setting and feedback obtained from stakeholders to refine the intervention. A mixture of qualitative and quantitative methods will be used in this project.

The trial hypothesises that the holistic, person-centred frailty-attuned intervention will benefit CHF patients not only in terms of improved physical function but also QoL and reduce hospitalisations. This might also reduce NHS costs associated with managing adverse outcomes of at-risk patients. On the wider level, the intervention could potentially improve the care and outcomes in patients with CHF nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 65 years or above.
  * Diagnosed with CHF for at least 1 year (Signs and symptoms of HF & either LVEF <40% or LVEF ≥40% with evidence of structural cardiac abnormality on echocardiogram including increased left atrial size, LV hypertrophy or impaired LV filling and/or raised natriuretic peptides: B-type natriuretic peptide (BNP) <35 pg/mL/ N-terminal pro-B-type natriuretic peptide (NT-proBNP) <125 pg/mL)
  * CFS ≥5
  * Willing to actively engage in a 12-week intervention developed by our team targeting older people with frailty and CHF
  * Willing to wear a wrist accelerometer for 7 days before the intervention as well as during the 12-week intervention to assess physical activity profile and monitor adherence to exercise programme
  * Willing to comply with all study requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study
  * Willing to provide feedback regarding the intervention in the form of interview/ focus groups/ surveys to help refine the intervention
  * Willing for audio recordings or note taking to take place during interviews/ focus groups

Exclusion Criteria:

* • Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study.

  * Significant cognitive impairment that affects the participant's ability to adhere to intervention.
  * Recent wrist fracture or operation that affects the participant's ability to wear a wrist accelerometer
  * Recent injury or operations that would significantly reduce the participants ability to engage in their normal daily activities
  * Participants who are currently recruited into another research study involving a lifestyle intervention
  * Participants who are undergoing major operations during the 12-week intervention
  * Participants unable to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults with frailty and chronic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Qualitative evaluation with stakeholders to identify gaps in current HF care pathway leading to unmet healthcare needs in older people living with frailty and CHF | Up to 6 months
  Obtained by focus groups and interviews with patients, carers and healthcare professionals.
Phase II: Co-design and production of a holistic, patient-centered intervention addressing various healthcare needs of older people living with frailty and CHF | Up to 6 months
  Obtained by focus groups and interviews with patients, carers and healthcare professionals.
Phase IIa: Time spent in sedentary, light, moderate and vigorous activity over monitoring duration | Up to 6 months
  Measured with accelerometer data.
Phase III: Change in physical function as assessed by the SPPB upon completion of 12-week intervention and at 6 month follow up (this may alter depending on findings from Phase II) | Up to 6 months
  Measured with Short Physical Performance Battery (SPPB) instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided